CLINICAL TRIAL: NCT01130285
Title: Validation of a Multi-gene Test for Lung Cancer Risk
Status: Active, not recruiting | Type: Observational
Sponsor: University of Toledo Health Science Campus (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Other Study IDs: UTHSC - 11; 1RC2CA148572-01 (NIH)
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Normal bronchial epithelial cell (NBEC) RNA. NBEC samples were obtained by bronchoscopic brushing after informed consent to this project was obtained. RNA was extracted and frozen in aliquots then archived. Two aliquots, were prepared for most subjects. In most cases, there were more than 1 microgram of RNA per aliquot.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Non-Lung Cancer, Heavy Smoker: Subjects will be ≥ 50 years of age and have a ≥ 20 pack year smoking history and will be either healthy volunteers or individuals undergoing diagnostic bronchoscopy, with absence of lung cancer documented at the time of enrollment.
  Interventions: Genetic: Lung Cancer Risk Test

INTERVENTIONS:
Genetic: Lung Cancer Risk Test — Measurement of gene expression in normal bronchial epithelial cells obtained at time of bronchoscopy.
  Other Names: LCRT

SUMMARY:
The purpose of this study is to determine the validity of a multi-gene Lung Cancer Risk Test (LCRT). In the process, the investigators will establish a bank of NBEC samples and corresponding blood samples from individuals demographically at increased risk for lung cancer.

DETAILED DESCRIPTION:
Because more than 160,000 individuals die of lung cancer/year in the United States alone, it is important to use the best possible methods to determine whether increased surveillance of individuals at highest risk for lung cancer will result in reduced lung cancer mortality. The Lung Cancer Risk Test (LCRT) proposed for evaluation promises to accurately identify the 10-15% of the population that is most susceptible to lung cancer based on genetic predisposition. More than 90 million individuals in the United States alone are demographically at high risk for lung cancer and potential candidates for increased surveillance.

ELIGIBILITY:
Inclusion Criteria:

* 20 or more pack year smoking history
* clinical need for diagnostic bronchoscopy or consent to study driven bronchoscopy

Exclusion Criteria:

* Lung Cancer within 3 months after the date of enrollment

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of subjects aged 50 to 90 and with 20 or more pack year smoking history, who are determined not to have lung cancer at the time of enrollment or within three months after the date of enrollment, and either a) volunteer for the study driven bronchoscopy, or b) have standard of care clinical need for diagnostic bronchoscopy (e.g. they may present with respiratory symptoms or abnormal test results consistent with the need for bronchoscopy).
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2011-05; Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Accuracy of LCRT to predict incidental lung cancer | from time of enrollment
  Time of diagnosis of incidental lung cancer will be compared to value of the investigational device, the Lung Cancer Risk Test (LCRT).

CONTACTS AND LOCATIONS:
Overall Officials: James Willey, MD, Principal Investigator — University of Toledo Health Science Campus
Locations (13):
- United States (13):
  - National Jewish Health, Denver, Colorado
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - University of Toledo, Health Science Campus, Toledo, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Tennessee Valley Veterans Admin., Nashville, Tennessee
  - Vanderbilt, Nashville, Tennessee
  - Inova Fairfax Hospital, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crawford EL, Levin A, Safi F, Lu M, Baugh A, Zhang X, Yeo J, Khuder SA, Boulos AM, Nana-Sinkam P, Massion PP, Arenberg DA, Midthun D, Mazzone PJ, Nathan SD, Wainz R, Silvestri G, Tita J, Willey JC. Lung cancer risk test trial: study design, participant baseline characteristics, bronchoscopy safety, and establishment of a biospecimen repository. BMC Pulm Med. 2016 Jan 22;16:16. doi: 10.1186/s12890-016-0178-4. PMID 26801409